CLINICAL TRIAL: NCT01475916
Title: Quality of Life in Asthmatic Children at School Age : Influence of Therapeutic Education
Brief Title: Quality of Life in Asthmatic Children at School Age
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: CHU-0105
Record Dates: First submitted 2011-09-23; First posted 2011-11-22 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Asthma
Keywords: Asthma; Educational program; Quality of life; School-aged children
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Educational program: consultation with paediatric pulmonologist — Longitudinal prospective study

SUMMARY:
Asthma is the most common chronic disease in childhood [1]. The advantage of an educational program in a global strategy of care has been established in asthma (decrease of nocturnal asthma, absence from work and school) [2, 3]. Therapeutic education of the patient permits the reduction of the rate of hospitalization, of the rate of emergencies visits and non-programmed visits. [3].

The WHO defines quality of life as an individual's perception of its place in existence, in the context of culture and value system in which he lives, in relation to its objectives, expectations, standards and concerns [4]. The basic point of this concept is the notion of perception, emphasizing the perspective of the person. It is a broad concept affected in a complex way by the subject's physical health, psychological state, level of independence, social relationships, and its relations with its environment. In the field of health, analyzing the quality of life includes objective aspects (living conditions, functional health) and subjective aspects (satisfaction, happiness, well-being) that allow to understand the situation of people in whole.

As defined by the WHO-Europe report published in 1996 [5], the therapeutic education aims to help patients acquire or maintain the competencies they need to best manage their lives with a chronic disease.

It is entirely part of the management of the patient. It includes organized activities designed to make patients aware and informed of their disease, of care organization and hospital procedures, and the behaviors related to health and disease. This is to help them and their families understand their illness and treatment, to work together and to gain autonomy from their disease in order to help maintain and improve their quality of life [6].

However, studies demonstrating the effectiveness of therapeutic patient education are still very few, especially in children. The need for prospective studies including the evaluation of the impact on quality of life was highlighted in a recent Cochrane meta-analysis [7]. It seems interesting for the authors to assess the improvement of the quality of life after educational sessions in children at school-age.

DETAILED DESCRIPTION:
Longitudinal prospective study

ELIGIBILITY:
Inclusion Criteria:

* School-aged (from 5 to 10 years old) asthmatic children consulting for the first time a paediatric pulmonologist

Exclusion Criteria:

* Other non-atopic chronic disease

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-04 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
AUQUEI questionnaire (Asthma Caregiver's Quality of Life) | 3 or 4 months after the diagnosis of asthma

SECONDARY OUTCOMES:
Clinical control of asthma measured by the Asthma Control Test | 3 or 4 months after the diagnosis of asthma
Frequence and severity of the exacerbations | 3 or 4 months after the diagnosis of asthma
assessment of pulmonary function by spirometry | 3 or 4 months after the diagnosis of asthma

CONTACTS AND LOCATIONS:
Overall Officials: André LABBE, Md, PhD, Principal Investigator — University Hospital, Clermont-Ferrand